CLINICAL TRIAL: NCT03552302
Title: Effects of Yoga Exercise on Tinnitus Handicap and Sleep Quality of the Participates With Tinnitus
Brief Title: Effects of Yoga Exercise on Participates With Tinnitus
Status: Completed | Type: Observational
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B10503015
Record Dates: First submitted 2017-02-07; First posted 2018-06-11 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2018-12

CONDITIONS: Tinnitus
Keywords: Yoga; Tinnitus; Sleep
MeSH Terms: conditions — Tinnitus | interventions — Yoga

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Yoga exercise for 12 weeks
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 1. Yoga stretch warm-up exercise for 15 minutes.
  2. Five kinds of yoga correction method for 30 minutes (abdominal breathing, throat breathing, wind box breathing, nasal alternating breathing, buzzing breathing).
  3. Great rest for 15 minutes

SUMMARY:
This study aimed to investigate the effectiveness of Yoga on the tinnitus handicap and sleep quality in humans. We selected adult participates with chronic tinnitus (>6 months). All participates performed Yoga exercise once per week at outpatient department under the guidance of a professional teacher, and performed once daily by themselves at home for 12 weeks. Questionnaires of Tinnitus Handicap Inventory and Pittsburgh Sleep Quality Index were measured before the start of this study, at the end of this study, and 1 month after the end of this study.

DETAILED DESCRIPTION:
Tinnitus is the auditory phantom sensation in the absence of external sound stimulation. Tinnitus that persisted more than six months without improvement can be called chronic tinnitus. One report proposed the neurophysiological model of tinnitus. In addition, tinnitus patients suffered from insomnia, irritability, anxiety and/or depression.

Current management of tinnitus is a drug-based treatment and/or nutritional supplementation. Music therapy, hearing aid therapy, and tinnitus retraining therapy (TRT), were also applied for patients with tinnitus. Even though, success rates of various tinnitus treatments were still unsatisfactory till now.

This study aimed to investigate the effectiveness of Yoga on the tinnitus handicap and sleep quality in humans. We selected adult participates with chronic tinnitus (>6 months). All participates performed Yoga exercise once per week at outpatient department under the guidance of a professional teacher, and performed once daily by themselves at home for 12 weeks. Questionnaires of Tinnitus Handicap Inventory and Pittsburgh Sleep Quality Index were measured before the start of this study, at the end of this study, and 1 month after the end of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participates with tinnitus persisted more than 6 months from ear, nose, and throat out-patient department.
2. No drug treatment for their tinnitus in recent 3 months.
3. No respiratory diseases (eg, asthma).
4. Normal cognitive function.
5. Normal language comprehension.

Exclusion Criteria:

1. Pregnant females or menopausal females with hormone replacement therapy.
2. Hypertension
3. Glaucoma.
4. Those who cannot express their opinions or follow orders.
5. Cancer patients.
6. Objective tinnitus.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Tinnitus participates.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from Assessment of the degree of tinnitus | 1. One week before yoga intervention. 2. Through study completion, an average of 12 week. 3. One month after the end of the study.
  Chinese version of Tinnitus Handicap Inventory (THI). There were 25 questions and totally 100 points in THI. The answer for each questions is classified into three levels (will, sometimes, will not), and answering "will" gave 4 points, answering "sometimes" gave 2 points, and answering "will not " gave 0 points. The higher the total scores, the more severe the tinnitus.

SECONDARY OUTCOMES:
Assessment of the degree of sleep quality. | 1. One week before yoga intervention. 2. Through study completion, an average of 12 week. 3. One month after the end of the study.
  Chinese version of Pittsburgh Sleep Quality Index (PSQI). There were 18 counted items and totally 21 points. The answer for each questions is classified into four levels (frequent, sometimes, rare, never), and answering "frequent" gave 3 points, answering "sometimes" gave 2 points, answering "rare" gave 1 point, and answering "never" gave 0 point. The higher the total scores, the more severe the sleep problem.

CONTACTS AND LOCATIONS:
Overall Officials: Juen-Haur Hwang, Ph. D., Study Chair — Dalin Tzu Chi General Hospital
Locations (1):
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No